CLINICAL TRIAL: NCT00132288
Title: A Randomized Controlled Trial Linking Clinical Quality Improvement Programs for Older Diabetics to a Community Based Activity Support Center
Brief Title: MY PALS: A Community-Based Physical Activity Support Program for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: James P. LoGerfo, MD, MPH, University of Washington Health Promotion Research Center
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 04-4349-E/A01
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2007-12-19 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus; Aging
Keywords: Aging; Frailty; Sedentary; Falls; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus; Frailty; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Motivational support — Participants in the PALS program at SE Seattle Senior Center are assigned a volunteer phone buddy who uses motivational interviewing techniques during bi weekly or monthly phone calls to encourage the participant to become more physically active.
  Other Names: Based on Stanford's Active Choices model.
Behavioral: PALS - Physical activity for lifetime success — Referral by a primary care provider to a community based support program to enhance uptake or maintenance of physical activity by the participants.

SUMMARY:
This is a study of whether physical activity of older adults can be improved by linking primary care clinics serving older adults to a community-based program that provides motivational support, including peer counselors, for engaging in and maintaining moderate levels of physical activity.

Health care providers at the participating study sites routinely assess and track diabetic patients' physical activity. In addition to this routine care, study volunteers are referred to a support program that has been modelled on the Active Choices Program. Changes in volunteers' levels of activity are measured at 3, 6, and 12 months.

DETAILED DESCRIPTION:
The MY PALS project will focus on developing an organized approach to increasing physical activity for clients who have already decided they are willing to increase activity or who might be having difficulty maintaining activity.

The MY PALS study will enroll consenting patients at clinics in Southeast Seattle-initially at two Puget Sound Neighborhood Health Center community clinics. These clinics have existing programs to provide better care for diabetic patients by encouraging and tracking physical activity, but the existing programs do not include community-based motivational supports.

Goals and objectives: The primary aim of My PALS is to determine the effectiveness of a support program to improve levels of physical activity in older diabetic patients in a diverse group of patients of clinics in SE Seattle. Secondary aims include: 1) identifying barriers to increased physical activity despite the offer or use of enhanced supports, and examining what those barriers imply for future study; and 2) estimating non-costs of the intervention.

The program consists of phone support, in-person counseling if the volunteer chooses, and access to a mentor if the volunteer chooses.

At initial contact, participants will complete a baseline questionnaire, including a the Seattle Rapid Assessment of Physical Activity (Seattle-RAPA). Participants desiring to meet in person with a peer counselor will discuss further plans for action and followup. In addition, participants who desire extra support will be offered the option of an ongoing peer mentor.

Participants will receive follow-up calls at the agreed upon intervals-usually no more than weekly, nor less than monthly for the first 3 months. At 3, 6 and 12 months, volunteers will again be asked to complete followup questionnaires. Copies of the plans and follow up activity scores will be sent to the volunteers' health care providers.

The primary outcome measure will be change in Seattle-RAPA score at 12 months in the intervention participants compared to the wait-listed control patients. The latter will be offered the intervention in Year 2.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 65 years and older. Depending on number of volunteers, may also include younger adults.
* English, Vietnamese, Tagalog, and Cambodian speakers.
* If successful, program will extend to non-diabetics older than 64 years

Exclusion Criteria:

* Cognitive impairment or mental illness precluding independent judgement
* Physician assessment that program is not appropriate, e.g., marked frailty

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2005-05; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in physical activity of those allocated to the intervention group compared to "wait-listed" controls as measured by the Seattle-Rapid Assessment of Physical Activity questionnaire | 1 year

SECONDARY OUTCOMES:
Change in level of activity for those contacted by community support program | 6 months
Change in activity level for those having a peer counselor | 6 months
Change in Hemoglobin A1c levels | 1 year
Determinants of choice in favor of study participation | does not apply

CONTACTS AND LOCATIONS:
Overall Officials: James LoGerfo, MD, Principal Investigator — University of Washington
Locations (1):
- Southeast Senior Center, Seattle, Washington, United States